CLINICAL TRIAL: NCT00587223
Title: A Prospective, Multicenter, Within Subject Controlled Study to Evaluate the Effect of Apligraf in Nonhealing Wounds of Subjects With Junctional or Dystrophic Epidermolysis Bullosa
Brief Title: Safety and Efficacy of Apligraf in Nonhealing Wounds of Subjects With Junctional or Dystrophic Epidermolysis Bullosa (EB)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient patient enrollment
Sponsor: Organogenesis (Industry)
Responsible Party: Katherine B. Giovino, Director of Clinical Operations, Organogenesis Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-EB-001-AG
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Epidermolysis Bullosa, Junctional; Epidermolysis Bullosa Dystrophica
MeSH Terms: conditions — Epidermolysis Bullosa, Junctional; Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Apligraf (a living bilayered cell therapy product)
  Interventions: Device: Apligraf
- 2 (Active Comparator): Dressing regimen comprised of a primary nonadherent dressing, nonstick gauze and standard dressing retainer.
  Interventions: Other: Standard dressing regimen

INTERVENTIONS:
Device: Apligraf — Up to 3 applications: Day 0, Month 1, Month 2.
  Arms: 1
Other: Standard dressing regimen — Dressing regimen will be comprised of a primary nonadherent dressing, nonstick gauze and standard dressing retainer
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the use of Apligraf for the treatment of nonhealing wounds in subjects with dystrophic or junctional epidermolysis bullosa. Apligraf will be evaluated for efficacy and safety compared to a conventional nonadherent dressing. A matched-pair design will be used to evaluate Apligraf treatment versus conventional treatment in 68 study pairs.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 2 and 65 years of age.
* Subject with clinical and histological diagnosis of junctional or dystrophic EB with documented electron microscopy or immunofluorescence microscopy.
* Subject has at least two non-adjacent EB lesions, at least 4 cm apart. The two selected EB lesions must be relatively matched in terms of diagnosis, location, level of erosion and size. Lesions may be on the same limb.
* Subject with dystrophic or junctional EB lesions between 10-44 cm2 present for at least 6 weeks. For the purposes of this study, a lesion is defined as a wound resulting from a post blister erosion.
* Subject who is a female of child-bearing potential (females >10 years of age) must have a documented negative urine or serum pregnancy test. Sexually active females must be practicing a medically proven form of contraception during the course of the study period.
* Subject or legal guardian must have read, understood and signed an institutional review board (IRB) approved Informed Consent Form or Assent Form.
* Subject and/or legal guardian must be able and willing to follow study procedures and instructions.

Exclusion Criteria:

* Subject with lesions only on the soles, posterior thigh or gluteus maximus.
* Subject whose lesion has healed 20% or greater in area from post debridement (if applicable) Baseline Screen (Visit 1) to post debridement Day 0 (Visit 2) as determined by wound tracings.
* Subject with uncontrolled diabetes mellitus (glycosylated HbA1C > 10%), cancer (biopsy confirmed active malignancy), or positive HIV test.
* Subject is a child (<18 years of age) who is currently receiving or has received oral steroid therapy exceeding a total daily dose of 0.5mg/kg for more than two weeks, radiation or other immuno-suppressive therapy which would interfere with wound healing within the past four weeks.
* Subject is an adult (>18 years of age) who is currently receiving or has received chronic high dose steroid therapy exceeding a total daily dose of 20mg for more than two weeks, radiation or other immuno-suppressive therapy which would interfere with wound healing within the past four weeks.
* Subject who is currently on or has received topical steroidal therapy within 30 days before screening. Inhaled steroids are allowed.
* Subject with the presence of acute infections in the areas intended for treatment.
* Subject with a history of squamous cell carcinoma.
* Known hypersensitivity to bovine collagen or to the components of the Apligraf agarose shipping medium.
* Subject who is lactating or pregnant (hCG positive as determined by lab testing).
* Subject is a child (<18 years of age) with liver (ALT/SGPT, ALP, AST/SGOT, bilirubin, total protein, LDH) and/or renal function (BUN and creatinine) tests > 2 x upper limit of normal (ULN). Albumin < 2.0 mg/dL.
* Subject is an adult (>18 years of age) with liver (ALT/SGPT, ALP, AST/SGOT, bilirubin, total protein, LDH) and/or renal function (BUN and creatinine) tests > 2 x upper limit of normal (ULN). Albumin < 2.0 mg/dL.
* Subject enrolled in any wound or investigational device study for any disease within the past four weeks.
* Subject who has received an investigational drug or biological treatment within three months.
* Subject previously treated with Apligraf, Dermagraft or any other cell therapy at the target sites.
* Subject with a history of alcohol or substance abuse within the previous year, which could interfere with study compliance such as inability to attend scheduled study visits or compliance with home dressing changes.
* Subject who, in the opinion of the investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Alvarez- Connelly, MD, Principal Investigator — University of Miami; Damien Bates, MD, PhD, FRACS (Plast.), Study Director — Organogenesis Inc.
Locations (5):
- United States (5):
  - Stanford University School of Medicine, Stanford, California
  - University of Miami - Miller School of Medicine, Miami, Florida
  - Columbia University Medical Center, New York, New York
  - Children's Hospital of Cincinnati, Cincinnati, Ohio
  - University of Texas, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from US hospital-based clinics. Recruitment was from December 2007 to December 2008.
Pre-assignment Details: A screening period of 1 week was utilized in the study design prior to randomization of study lesions to Apligraf or control at Day 0.
Groups:
- Apligraf: Within subject control: 2 lesions per subjects randomized to receive Apligraf or Control treatment. The lesion treated with Apligraf receives a single topical application of Apligraf to cover the lesion.
Period: Overall Study
Arm/Group | Apligraf
Started | 1 (Study design was within-subject control. Only 1 subject was enrolled in the study.)
Completed | 0 (Subject withdrawn from study at Day 7.)
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Apligraf/Control: Apligraf (a living bilayered cell therapy product) Control (a primary nonadherent dressing, nonstick gauze, retainer dressing)
Arm/Group | Apligraf/Control
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Wounds First Achieving 100% Epithelialization of Tissue With the Absence of Drainage (i.e. Complete Wound Closure) Through Study Week 12
Time Frame: Through 12 weeks
Population: no analysis performed as only 1 subject enrolled
Measure: Number; unit: proportion (%) of treated wounds
Groups:
- Control: Within subject control: 2 lesions per subject randomized to receive Apligraf or Control treatment. Control treated lesion receives standard wound dressings.
Arm/Group | Apligraf | Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time Until Complete Closure
Time Frame: through 12 weeks
Population: no analysis performed as only 1 subject enrolled
Measure: Number; unit: days
Groups:
- Control: Within subject control: 2 lesions per subject randomized to receive Apligraf or Control treatment. Control treated lesions receive standard wound dressings.
Arm/Group | Apligraf | Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Rate of Complete Wound Closure Over Time
Time Frame: through 12 weeks
Population: no analysis performed as only 1 subject enrolled
Measure: Number; unit: change in area from baseline to Week 12
Groups:
- Control: Within subject control: 2 lesions per subjects randomized to receive Apligraf or Control treatment. Control lesions are treated with standard wound dressings.
Arm/Group | Apligraf | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Recurrence of Epidermolysis Bullosa (EB) Lesions
Time Frame: through 12 months
Population: no analysis performed as only 1 subject enrolled
Measure: Number; unit: proportion (%) of treated wounds
Arm/Group | Apligraf | Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Reduction of Intensity of Pain
Time Frame: through 12 weeks
Population: no analysis performed as only 1 subject enrolled
Measure: Number; unit: change in pain intensity between groups
Arm/Group | Apligraf | Control
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Proportion of Wounds Experiencing an Adverse Event
Time Frame: through 12 months
Population: There was only 1 enrolled subject in the study; this endpoint was descriptively reported, no statistical analyses were performed.
Measure: Number; unit: proportion of treated wounds
Arm/Group | Apligraf | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: December 2007 through August 2008
Arm/Group | Apligraf
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apligraf (N=1)
Fever (General disorders) | 1 (1)
Wound Infection (signs and symptoms) (Infections and infestations) | 1 (2) — Two events reported, both treated lesions were simulataneously reported as having a wound infection.

LIMITATIONS AND CAVEATS:
Study terminated early, the 1 enrolled subject subsequently discontinued study at Day 7.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before publishing PI shall submit copies of any proposed publication/presentation to Sponsor for review at least 30 days in advance of submission. Sponsor shall review the data provided in proposed publication against the Study database for consistency. Sponsor reserves right to delete any Confidential Information/proprietary information of Sponsor from the proposed publication/presentation. Sponsor may extend such review period for another 90 days.